CLINICAL TRIAL: NCT05942963
Title: PEARL-DM: Efficacy of Empagliflozin and Pioglitazone in Diabetic Patients With NAFLD; Randomized Controlled Trial From Pakistan.
Brief Title: Efficacy of Empagliflozin and Pioglitazone in Diabetic Patients With NAFLD
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jinnah Postgraduate Medical Centre (Other Government)
Responsible Party: Principal Investigator, ZA, Associate professor, Jinnah Postgraduate Medical Centre
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: JSMU/IRB/2023/709
Record Dates: First submitted 2023-06-16; First posted 2023-07-12 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-07

CONDITIONS: Non-Alcoholic Fatty Liver Disease; Type2diabetes
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — empagliflozin; Pioglitazone; Metformin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group A (Experimental): SOC+ Empagliflozin + Pioglitazone
  Interventions: Drug: Empagliflozin 10 MG; Drug: Pioglitazone 15mg; Drug: Metformin
- Group B (Experimental): SOC +Empagliflozin
  Interventions: Drug: Empagliflozin 10 MG; Drug: Metformin
- Group C (Experimental): SOC+ Pioglitazone
  Interventions: Drug: Pioglitazone 15mg; Drug: Metformin
- Group D (Active Comparator): SOC only
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Empagliflozin 10 MG — 10-25 mg/day
  Arms: Group A; Group B
Drug: Pioglitazone 15mg — 15-45 mg/day
  Arms: Group A; Group C
Drug: Metformin — 1000mg-2850mg/ day

SUMMARY:
This clinical trial will yield results about the therapeutic effect of combining pioglitazone with SGLT2i in people suffering from NAFLD associated with T2DM. Study participants will be asked to fill out a few questions on proforma that will obtain demographic information as well as information relating to their health. In addition, some blood tests will be done following standard procedures.

DETAILED DESCRIPTION:
This is a randomized clinical trial conducted to compare the efficacies of pioglitazone and empagliflozin in people suffering from NAFLD associated with T2DM.

Randomization will be done using card randomization. Four different color-coded cards will be kept. Any card will be randomly picked for the patient fulfilling inclusion criteria and will be treated according to the allocated treatment arm mentioned on the card

Written informed consent will be obtained from the immediate attendant of the patient. All ethical considerations will be followed.

Our research has been approved by Jinnah Sindh Medical University, Karachi. For this approval, the investigators have made every effort to ensure the confidentiality of research data collected from all our participants in this survey. The information collected will be stored with the investigators only in the form of de-identified information and will be retained in a secure place under lock and key. Any results that will be generated will be presented on a collective basis, and will not contain the participants name or any other personal details.

Data entry and analysis will be done using SPSS Software version 23. Study analysis will be done using the principle of intention to treat. The mean scores will be compared pre and post-intervention using paired t-test. The association of age, gender, and grade of fatty liver will be compared with different groups using correlation and regression models. All analyses will be at a confidence Interval of 95% and a p-value <.05.

ELIGIBILITY:
Inclusion Criteria:

* T2DM patients with NAFLD glycated
* APRI scores of more than 1.5

Exclusion Criteria:

* Patients having type 1 diabetes
* evidence of advanced/decompensated cirrhosis (on the basis of a Child-Pugh score of more than 7 and MELD of more than 15)
* hepatocellular carcinoma (evidence on ultrasound or alpha-fetoprotein)
* patient suffering from acute or chronic hepatitis
* biliary disease
* HIV
* hemochromatosis
* autoimmune conditions (alpha-1 antitrypsin deficiency, autoimmune hepatitis, Wilson's disease)
* renal dysfunction with GFR [eGFR] <30 mL/min/1.73m2
* history of alcohol ( male >30 g/d and female;20 g/d)
* history of cancer or undergoing treatment for cancer,
* use of amiodarone, tamoxifen, sodium valproate, corticosteroids, methotrexate, ursodeoxycholic acid, S-adenosyl methionine, betaine, silymarin, gemfibrozil
* using supplements including vitamin E, vitamin C, zinc, and selenium or antioxidant agents over the last 3 months
* history of cardiovascular events within the past 3 months
* pregnancy or breastfeeding
* contraindications to empagliflozin use (history of recurrent urogenital infections, current or previous gangrene, or hypersensitivity reaction to the molecule)
* history of bladder cancer
* morbid obesity (BMI greater than 35).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2023-10 (Estimated); Primary Completion 2024-04 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
A change in liver steatosis will be assessed through fibro CAP score. | Will be assessed at enrollment.
  Fibro-controlled attenuation parameter (fibro CAP). The parameter range is commonly between 100 and 400 dB/m, and the greater the reading worse will be the outcome.
A change in liver steatosis will be assessed through fibro CAP score. | Will be assessed at 168th day post enrollment.
  Fibro-controlled attenuation parameter (fibro CAP). The parameter range is commonly between 100 and 400 dB/m, and the greater the reading worse will be the outcome.

SECONDARY OUTCOMES:
change in SF-36 scores | Quality of life will be assessed 84th day post enrollment.
  36-Item Short Form Survey (SF-36) assesses eight health concepts: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions. A higher score defines a more favorable health state.
change in SF-36 scores | Quality of life will be assessed at day 252 post enrollment.
  36-Item Short Form Survey (SF-36) assesses eight health concepts: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions. A higher score defines a more favorable health state.
change in liver fibrosis will be assessed through the FIB-4 index. | at enrollment.
  Fibrosis-4 index (FIB-4). Low scores will indicate better outcomes (less fibrosis).
change in liver fibrosis will be assessed through the FIB-4 index. | 84th day post enrollment.
  Fibrosis-4 index (FIB-4). Low scores will indicate better outcomes (less fibrosis).
change in liver fibrosis will be assessed through the FIB-4 index. | at 168th day post enrollment.
  Fibrosis-4 index (FIB-4). Low scores will indicate better outcomes (less fibrosis).
change in liver fibrosis will be assessed through the FIB-4 index. | at day 252 post enrollment.
  Fibrosis-4 index (FIB-4). Low scores will indicate better outcomes (less fibrosis).
change in liver fibrosis will be assessed through the APRI Score | at enrollment.
  AST to platelet ratio index (APRI) Score. Lower the value better the outcome (less fibrosis)
change in liver fibrosis will be assessed through the APRI Score | 84th day post enrollment.
  AST to platelet ratio index (APRI) Score. Lower the value better the outcome (less fibrosis)
change in liver fibrosis will be assessed through the APRI Score | at 168th day post enrollment.
  AST to platelet ratio index (APRI) Score. Lower the value better the outcome (less fibrosis)
change in liver fibrosis will be assessed through the APRI Score. | at day 252 post enrollment.
  AST to platelet ratio index (APRI) Score. Lower the value better the outcome (less fibrosis)
change in liver fibrosis will be assessed through the NFS Score. | at enrollment.
  NAFLD fibrosis score (NFS). Lower the value better the outcome (less fibrosis)
change in liver fibrosis will be assessed through the NFS Score. | at 84th day post enrollment.
  NAFLD fibrosis score (NFS). Lower the value better the outcome (less fibrosis)
change in liver fibrosis will be assessed through the NFS Score. | at 168th day post enrollment.
  NAFLD fibrosis score (NFS). Lower the value better the outcome (less fibrosis)
change in liver fibrosis will be assessed through the NFS Score. | at day 252 post enrollment.
  NAFLD fibrosis score (NFS). Lower the value better the outcome (less fibrosis)
Change in hepatic steatosis through the FLI score. | at enrollment.
  Fatty liver index (FLI). Lower the value better the outcome
Change in hepatic steatosis through the FLI score. | at 84th day post enrollment.
  Fatty liver index (FLI). Lower the value better the outcome
Change in hepatic steatosis through the FLI score. | at 168th day post enrollment.
  Fatty liver index (FLI). Lower the value better the outcome
Change in hepatic steatosis through the FLI score. | at day 252 post enrollment.
  Fatty liver index (FLI). Lower the value better the outcome
Change in Insulin resistance will be assessed through HOMA-2IR/IR scale. | at enrollment.
  homeostatic model assessment-2IR (HOMA-2IR/IR). The lower the value better the outcome.
Change in Insulin resistance will be assessed through HOMA-2IR/IR scale. | at 84th day post enrollment.
  homeostatic model assessment-2IR (HOMA-2IR/IR). The lower the value better the outcome.
Change in Insulin resistance will be assessed through HOMA-2IR/IR scale. | at 168th day post enrollment.
  homeostatic model assessment-2IR (HOMA-2IR/IR). The lower the value better the outcome
Change in Insulin resistance will be assessed through HOMA-2IR/IR scale. | at day 252 post enrollment.
  homeostatic model assessment-2IR (HOMA-2IR/IR). The lower the value better the outcome.
Change in the LFT. | At enrollment.
  Liver Function test (LFT) such as alanine transaminase, aspartate transaminase, bilirubin, albumin, alkaline phosphatase, gamma-glutamyl transferase .
Change in the LFT. | 84th day post enrollment.
  Liver Function test (LFT) such as alanine transaminase, aspartate transaminase, bilirubin, albumin, alkaline phosphatase, gamma-glutamyl transferase .
Change in the LFT. | at 168th day post enrollment.
  Liver Function test (LFT) such as alanine transaminase, aspartate transaminase, bilirubin, albumin, alkaline phosphatase, gamma-glutamyl transferase .
Change in the LFT. | at day 252 post enrollment.
  Liver Function test (LFT) such as alanine transaminase, aspartate transaminase, bilirubin, albumin, alkaline phosphatase, gamma-glutamyl transferase .
Change in weight | at enrollment.
  weight. lower the levels better the outcome.
Change in weight | at 84th day post enrollment.
  weight. lower the levels better the outcome.
Change in weight | at 168th day post enrollment.
  weight. lower the levels better the outcome.
Change in weight | at day 252 post enrollment.
  weight. lower the levels better the outcome.
Change in random blood sugar | at enrollment.
  random blood sugar
Change in random blood sugar | at 84th day post enrollment.
  random blood sugar.
Change in random blood sugar | at 168th day post enrollment.
  random blood sugar.
Change in random blood sugar | at day 252 post enrollment.
  random blood sugar. lower the levels better the outcome.
Change in waist circumference | at enrollment.
  waist circumference. lower the levels better the outcome.
Change in waist circumference | at 84th day post enrollment.
  waist circumference. lower the levels better the outcome.
Change in waist circumference | at 168th day post enrollment.
  waist circumference. lower the levels better the outcome.
Change in waist circumference | at day 252 post enrollment.
  waist circumference. lower the levels better the outcome.
Change in HbA1c | at enrollment.
  hemoglobin A1c (HbA1c).lower the levels better the outcome.
Change in HbA1c | at 84th day post enrollment.
  hemoglobin A1c (HbA1c).lower the levels better the outcome.
Change in HbA1c | at 168th day post enrollment.
  hemoglobin A1c (HbA1c).lower the levels better the outcome.
Change in HbA1c | at day 252 post enrollment.
  hemoglobin A1c (HbA1c).lower the levels better the outcome.
Change in Body mass index | at enrollment.
  Body mass index. lower the levels better the outcome.
Change in body mass index | at 84th day post enrollment.
  body mass index. lower the levels better the outcome.
Change in body mass index | at 168th day post enrollment.
  body mass index. lower the levels better the outcome.
Change in body mass index | at day 252 post enrollment.
  body mass index. lower the levels better the outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical ICU, Jinnah Postgraduate Medical Centre, Karachi, Sindh, Pakistan